CLINICAL TRIAL: NCT05543096
Title: A Retrospective PMCF Study Evaluating the Safety and Clinical Performance of the Adroit Guiding Catheter, the Cordis Transradial Access Devices (RAIN Sheath and Avanti Plus Transradial Kit), the Cordis Diagnostic Catheters (Super Torque, Super Torque MB, Super Torque Plus, Infiniti 4F, Infiniti 5F/6F, Tempo 4F, Tempo Aqua, High Flow and Pigtail Straightener) and the Cordis Guidewires (ATW, Stabilizer and Wizdom) for Percutaneous Coronary Interventions.
Brief Title: PMCF Study for Cardiology Access Procedures
Status: Completed | Type: Observational
Sponsor: Cordis US Corp. (Industry)
Collaborators: FCRE (Foundation for Cardiovascular Research and Education) (Other)
Responsible Party: Sponsor
Other Study IDs: FCRE-220111_Cardio
Record Dates: First submitted 2022-06-29; First posted 2022-09-16 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Coronary Artery Disease
Keywords: Cardiology
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Adroit Guiding Catheter, Cordis Transradial Access Devices, Cordis Diagnostic Catheters, Cordis Guidewires — Observation

SUMMARY:
This Post-market clinical follow-up (PMCF) study is designed as retrospective, multi-center study to collect real-life data.

A multi-center design is used to ensure a representative sample of the physicians who have performed the procedure and to provide a reasonable enrolment period for the required data to be collected.

The rationale of this study is to confirm and support the clinical safety and performance of any of these products in a real-word population of 200 patients who underwent an endovascular intervention within standard-of-care (SOC) where at least 1 of the products (named above) from Cordis US Corp were used.

DETAILED DESCRIPTION:
Treatment of coronary artery disease (CAD) is dependent on percutaneous coronary intervention (PCI). PCI includes a group of minimally invasive (non-surgical) procedures to treat narrowing of the coronary arteries and therefore restore arterial blood flow. PCI techniques have significantly improved over time1 and requires cardiac catherterization and an experienced physician. In the field of catheters, there are a variety of options from Diagnostic Catheters, Guiding Catheters, Guidewires or even Transradial Acces Devices1-5.

All devices have different advantages and disadvantages and an appropriate selection is a requirement for successful angioplasty of coronary artery lesions2,3. Which device to choose depends on the anatomy of the vessel, the type of lesion and the technique used for the treatment. The different Catheters and Access Devices (Diagnostic Catheters, Guiding Catheters, Guidewires and Transradial Acces Devices) have proven their functionality and safety over the years and have become widely accepted supportive devices for the treatment of coronary atery disease. For example, the technical sucess for Diagnostic Catheters is high with about 95% technical success and about 100% procedural succes6-17.

In this regard, the purpose of the current post market surveillance trial is to assess the safety and efficacy of different devices from Cordis (Adroit Guiding Catheter, Cordis Transradial Access Devices, Cordis Diagnostic Cathheters, and Cordis Guidewires). The devices under investigation in the current study are the Adroit Guiding Catheter, Cordis Transradial Access Devices (RAIN Sheath and Avanti Plus Transradial Kit), Cordis Diagnostic Cathheters (Super Torque, Super Torque MB, Super Torque Plus, Infiniti 4F, Infiniti 5F/6F, Tempo 4F, Tempo Aqua, High Flow and Pigtail Straightener), Cordis Guidewires (ATW, Stabilizer, Wizdom), which are described in detail in section 3.1.

ELIGIBILITY:
Inclusion Criteria:

1. Corresponding to the CE-mark indications/contra-indications and according to the current medical guidelines for percutaneous coronary intervention (PCI).
2. Patient is >18 years old at the conduction of the procedure.
3. Patient is eligible for treatment with Adroit Guiding Catheter Cordis Transradial Access Devices

   * RAIN Sheath
   * Avanti Plus Transradial Kit Cordis Diagnostic Cathheters
   * Super Torque
   * Super Torque MB
   * Super Torque Plus
   * Infiniti 4F
   * Infiniti 5F/6F
   * Tempo 4F
   * Tempo Aqua
   * High Flow
   * Pigtail Straightener Cordis Guidewires
   * ATW
   * Stabilizer
   * Wizdom as described in the IFU for each device.

Exclusion Criteria:

1. Anatomy or size of vessels that did not allow appropriate usage of the study devices, following IFU of the study devices.
2. Known contraindication and/or allergy to (a component of) an study device as described in the IFU of the devices.
3. Women who were pregnant or lactating at the time of the procedure.
4. Any patient who was hemodynamically unstable at onset of procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diseased patients with CAD who underwent a PCI within standard-of-care (SOC) of the coronary arterial vessel. In this PMCF minimally invasive medical devices will be used. Indications for which the study devices are intended are listed in section 3.1. Patients will be selected based on the investigator's assessment and evaluation of the underlying disease retrospective. The patient's medical condition should have been stable, with no underlying medical condition which would prevent them from undergoing the required endovascular intervention at the time of procedure.
  The total sample size for this PMCF study is 200 patients, divided over up to 20 sites, throughout an enrolment period of 6 months.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2022-05-23 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-09-07 (Actual)

PRIMARY OUTCOMES:
Primary Safety Endpoint: Freedom from Serious Adverse Events and Serious Adverse Device Effects | 30 days after procedure
  Freedom from SAEs and SADEs during the procedure and up to 30 days after the procedure
Primary Efficacy Endpoint: Successful crossing, instroduction and deployment | 30 days post procedure
  Technical success rate defined as successful crossing, instroduction and deployment of Adroit Guiding Catheter according to the IFU and without device related deficiencies
Primary Efficacy Endpoint: Successful crossing, instroduction and deployment | 30 days post procedure
  Technical success rate defined as successful crossing, instroduction and deployment of Cordis Transradial Access Device RAIN Sheath according to the IFU and without device related deficiencies
Primary Efficacy Endpoint: Successful crossing, instroduction and deployment | 30 days post procedure
  Technical success rate defined as successful crossing, instroduction and deployment of Cordis Transradial Access Device Avanti Plus Transradial Kit according to the IFU and without device related deficiencies
Primary Efficacy Endpoint: Successful crossing, instroduction and deployment | 30 days post procedure
  Technical success rate defined as successful crossing, instroduction and deployment of Cordis Diagnostic Cathheter Super Torque according to the IFU and without device related deficiencies
Primary Efficacy Endpoint: Successful crossing, instroduction and deployment | 30 days post procedure
  Technical success rate defined as successful crossing, instroduction and deployment of Cordis Diagnostic Cathheter Super Torque MB according to the IFU and without device related deficiencies
Primary Efficacy Endpoint: Successful crossing, instroduction and deployment | 30 days post procedure
  Technical success rate defined as successful crossing, instroduction and deployment of Cordis Diagnostic Cathheter Super Torque Plus according to the IFU and without device related deficiencies
Primary Efficacy Endpoint: Successful crossing, instroduction and deployment | 30 days post procedure
  Technical success rate defined as successful crossing, instroduction and deployment of Cordis Diagnostic Cathheter Infiniti 4F according to the IFU and without device related deficiencies
Primary Efficacy Endpoint: Successful crossing, instroduction and deployment | 30 days post procedure
  Technical success rate defined as successful crossing, instroduction and deployment of Cordis Diagnostic Cathheter Infiniti 5F/6F according to the IFU and without device related deficiencies
Primary Efficacy Endpoint: Successful crossing, instroduction and deployment | 30 days post procedure
  Technical success rate defined as successful crossing, instroduction and deployment of Cordis Diagnostic Cathheter Tempo 4F according to the IFU and without device related deficiencies
Primary Efficacy Endpoint: Successful crossing, instroduction and deployment | 30 days post procedure
  Technical success rate defined as successful crossing, instroduction and deployment of Cordis Diagnostic Cathheter Tempo Aqua according to the IFU and without device related deficiencies
Primary Efficacy Endpoint: Successful crossing, instroduction and deployment | 30 days post procedure
  Technical success rate defined as successful crossing, instroduction and deployment of Cordis Diagnostic Cathheter High FLow according to the IFU and without device related deficiencies
Primary Efficacy Endpoint: Successful crossing, instroduction and deployment | 30 days post procedure
  Technical success rate defined as successful crossing, instroduction and deployment of Cordis Diagnostic Cathheter Pigtail Straightener according to the IFU and without device related deficiencies
Primary Efficacy Endpoint: Successful crossing, instroduction and deployment | 30 days post procedure
  Technical success rate defined as successful crossing, instroduction and deployment of Cordis Guidewire ATW according to the IFU and without device related deficiencies
Primary Efficacy Endpoint: Successful crossing, instroduction and deployment | 30 days post procedure
  Technical success rate defined as successful crossing, instroduction and deployment of Cordis Guidewire Stabilizer according to the IFU and without device related deficiencies
Primary Efficacy Endpoint: Successful crossing, instroduction and deployment | 30 days post procedure
  Technical success rate defined as successful crossing, instroduction and deployment of Cordis Guidewire Wizdom according to the IFU and without device related deficiencies

SECONDARY OUTCOMES:
Secondary Efficacy Endpoint: Successful crossing, introduction and deployment | 30 days post procedure
  Technical success rate defined as successful crossing, introduction and deployment of Vista Brite Tip Guiding Catheter according to the respective IFU and without device related deficiencies
Secondary Efficacy Endpoint: Successful crossing, introduction and deployment | 30 days post procedure
  Technical success rate defined as successful crossing, introduction and deployment of Cordis vascular access device RAILWAY Shealthless Access System according to the respective IFU and without device related deficiencies
Secondary Efficacy Endpoint: Successful crossing, introduction and deployment | 30 days post procedure
  Technical success rate defined as successful crossing, introduction and deployment of Cordis vascular access device Avanti+ according to the respective IFU and without device related deficiencies
Secondary Efficacy Endpoint: Successful crossing, introduction and deployment | 30 days post procedure
  Technical success rate defined as successful crossing, introduction and deployment of Cordis vascular access device Brite - Tip according to the respective IFU and without device related deficiencies
Secondary Efficacy Endpoint: Successful crossing, introduction and deployment | 30 days post procedure
  Technical success rate defined as successful crossing, introduction and deployment of Cordis vascular access device Vista Brite IG according to the respective IFU and without device related deficiencies
Secondary Efficacy Endpoint: Successful crossing, introduction and deployment | 30 days post procedure
  Technical success rate defined as successful crossing, introduction and deployment of Cordis vascular access device Vessel Dilator according to the respective IFU and without device related deficiencies
Secondary Efficacy Endpoint: Successful crossing, introduction and deployment | 30 days post procedure
  Technical success rate defined as successful crossing, introduction and deployment of Cordis vascular closure device MynxGrip according to the respective IFU and without device related deficiencies
Secondary Efficacy Endpoint: Successful crossing, introduction and deployment | 30 days post procedure
  Technical success rate defined as successful crossing, introduction and deployment of Cordis vascular closure device Mynx Control according to the respective IFU and without device related deficiencies
Secondary Efficacy Endpoint: Successful crossing, introduction and deployment | 30 days post procedure
  Technical success rate defined as successful crossing, introduction and deployment of Cordis Guidewire Emerald according to the respective IFU and without device related deficiencies.

CONTACTS AND LOCATIONS:
Locations (8):
- Austria (6):
  - Kepler Universitätsklinikum GmbH, Linz
  - Ordensklinikum Linz GmbH, Linz
  - ST. Poelten, Sankt Pölten
  - Klinik Favoriten, Vienna
  - Klinik Floridsdorf, Vienna
  - Klinikum Wels Grieskirchen, Wels
- Belgium (2):
  - VZW Jessa Ziekenhus, Hasselt
  - AZ Sint Nikolaas, Sint-Niklaas

IPD SHARING:
Plan to Share IPD: Undecided